CLINICAL TRIAL: NCT02850562
Title: Diet and Exercise Interventions to Increase Muscle Strength and Function:A Randomized Controlled Trial
Brief Title: Diet and Exercise Interventions to Increase Muscle Strength and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Responsible Party: Principal Investigator, Bonny Specker, Professor, South Dakota State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-1607001-EXP
Record Dates: First submitted 2016-07-21; First posted 2016-08-01 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Sarcopenia; Metabolic Syndrome X
Keywords: body composition,; Dual-Energy X-Ray Absorptiometry; sarcopenia; peripheral quantitative computed tomography; muscle density; elderly
MeSH Terms: conditions — Obesity; Sarcopenia; Metabolic Syndrome | interventions — Walking; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walking (Active Comparator): The Walking Arm will walk 5 times per week for at least 10 minutes/day at the start of the study and build to 30 minutes/day by the 3-month time point.
  Interventions: Behavioral: Walking
- Walking + Exercise (Experimental): The Walking + Exercise Arm will walk 2 times per week for at least 10 minutes/day at the start of the study and build to 30 minutes/day by the 3-month time point and in addition, complete exercises to improve strength and balance on 3 days each week.
  Interventions: Behavioral: Walking + Exercise

INTERVENTIONS:
Behavioral: Walking — The Walking Arm will walk 5 times per week for at least 10 minutes/day at the start of the study and build to 30 minutes/day by the 3-month time point.
  Other Names: Control
  Arms: Walking
Behavioral: Walking + Exercise — The Walking + Exercise Arm will walk 2 times per week for at least 10 minutes/day at the start of the study and build to 30 minutes/day by the 3-month time point and in addition, complete exercises to improve strength and balance on 3 days each week.
  Other Names: Exercise
  Arms: Walking + Exercise

SUMMARY:
The objective of this study is to test the effects of a healthy diet & walking (Controls) compared to a healthy diet, walking, and balance/strength exercises (Intervention) on muscle density in two populations: elderly individuals and obese individuals. The intervention will be 3 months in length. During this time, both Control and Intervention groups will meet one time each week for educational sessions on healthy diet strategies and to participate in a group walk for the Control group or group exercises for the Intervention group. The Control group will be asked to walk on their own an additional 4 times per week (5 times total) for at least 10 minutes/day at the start of the study and build to 30 minutes/day by the 3-month time point. The Intervention group will walk two times per week using the same criteria as above, and in addition will do balance/strength exercises on a total of three days per week. Measurements will be made at baseline, at intervention completion (3 months) and at a follow-up (6 months -3 months after completion of the intervention). At 3 months, the control group will be invited to add the balance/strength exercises.

The hypotheses are that adding balance & strength exercises to a healthy diet plan will increase muscle density (decrease fat infiltration) and improve muscle function in the elderly and in the obese populations. Increases in muscle density are expected to show greater improvements in muscle function in the elderly population, while it is speculated that greater improvements in metabolic measures will show in the obese population. Participants in the intervention group will have a greater reduction in falls and less hospital, ER & clinic visits compared to the control group, but both groups will have an improved quality of life, positive changes in eating behaviors, and decreased perceived stress.

DETAILED DESCRIPTION:
Sarcopenia, the loss of skeletal lean mass and muscle strength, occurs in elderly but also may be present in obese individuals due fat infiltration of the muscle. Loss of lean mass along with fat infiltration into skeletal muscle causes decreased muscle density, which contributes to decline in muscle function. Increases in muscle density are expected to improve muscle function as well as metabolic function. This study will test the effects of a healthy diet & walking (Controls) compared to a healthy diet, walking, and balance/strength exercises (Intervention) on muscle density in two populations: elderly individuals and obese individuals. The intervention will be 3 months in length. The Control group will walk 5 times per week for at least 10 minutes/day at the start of the study and build to 30 minutes/day by the 3-month time point. The Intervention group will walk two times per week using the same criteria, and in addition will do balance/strength exercises on three days per week. At 3 months, the control group will be invited to add the balance/strength exercises.

Study visits at baseline, at intervention completion (3 months), and at a follow-up (6 months -3 months after completion of the intervention) will include: questionnaires; anthropometric measures, body composition, muscle density and trabecular bone measures; muscle function and strength testing; activity measures; diet recall; metabolic measures (waist circumference, blood pressure, fasting blood sugar, triglyceride, HDL cholesterol); and erythrocyte sedimentation rate (see Outcome Measures below for detailed measures).

Healthy Diet Education Sessions: USDA's MyPlate, was introduced in 2010, as the new guidelines for proper dietary nutrition. These guidelines, developed by the USDA in conjunction with the Department of Health and Human Services are designed to serve as the "cornerstone of Federal nutrition policy and nutrition education activities" (USDA Dietary Guidelines, 2011). Each week participants will attend a healthy diet education session based on MyPlate Dietary Guidelines. Dr. Holm will oversee the lessons that will be developed and implemented by SDSU Health and Nutritional Sciences students. Twelve lessons will be given and cycled over 3 month periods so that no matter when a participant enters the study, the same twelve sessions will be completed as they go through the study program. Focus of the sessions will be on topics such as portion size, reading food labels, calorie intake and burning, tips for grocery shopping, healthy recipes, food groups, healthy fats, carbohydrates and proteins, etc. Each lesson will take approximately 20 minutes with a group activity session to follow.

Exercise Interventions:

Control Group - The exercise intervention for the control group is walking. Walking will be expected to be completed 5 days per week and done at the participant's physical ability/pace. At the start of the study, the participant will complete at least 10 minutes per day or more according to their physical ability. By the end of the study, this is expected to increase to 30 minutes of walking each day and can be completed in 10-minute intervals throughout the day. One day per week, the control group participants will be invited to do a 'group walk' that will be on the same day of the week following the dietary education lesson. Participants will keep weekly walking logs to record the time they walk each day for the purpose of exercise, not as part of daily activities. Weekly logs will be collected and a new one issued each week during the dietary education lesson. Exercise compliance will be calculated using these logs.

Intervention Group - The intervention group will walk as described above, but only on two days per week. Three days per week, exercises focusing on strength and balance will completed (see Five Esslinger Exercises for Strength and Balance below). These exercises can be completed in one bout, or spread throughout the day. Participants will be given weekly logs to record their walking and exercise activities similar to the control group as described above. Participants will be instructed by study personnel including South Dakota State University Health and Nutritional Science students on how to properly do the exercises to their level of ability with a focus on modifications to ensure safety and prevent injuries or falls. One day per week, the intervention group will be invited to do a 'group exercise session' following the dietary education lesson. South Dakota State University Health and Nutritional Science students will assist in teaching the proper form and safety measured to perform the exercises and assist with the group sessions.

ELIGIBILITY:
Inclusion Criteria:

Two population groups will be recruited:

1. Women and Men > 18 years of age and < 70 years of age who have a BMI >35.
2. Women and Men 70 years of age or older.

Exclusion Criteria:

* Women and men younger than 18 years of age will be excluded.
* Women and men aged > 18 years and < 70 years with a BMI < 35 kg/m2 will be excluded.
* Women and men with the following conditions will be excluded unless given permission by their doctor: Taking medications for heart conditions or high blood pressure; chest pain with our without physical activity; loss of balance or dizziness; bone or joint problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Density | Change from Baseline to 3 Months, Change from Baseline to 6 Months
  Muscle density measures will be obtained by peripheral quantitative computed tomography (pQCT) using the XCT3000 densitometer (Orthometrix, Inc.). The image is obtained while the participant is seated and the right leg is extended through the gantry of the device. A scout view will be obtained to reference the end of the tibia and a slice at 66% of the tibia length from the distal end will be obtained. The 66% site is the thickest part of the calf and is used to measure muscle density in mg/cm3. The imaging will take approximately 10 minutes and the total radiation effective dose for the scout view and two slices is considered low (< 1 μSv). The change in muscle density in mg/cm3 from baseline to intervention completion (3 months) will be used to test the effect of the intervention. The change in muscle density in mg/cm3 from baseline to follow-up (6 months) will be used to test the persistent effect of the intervention.
Change in Calf Muscle Peak Torque | Change from Baseline to 3 Months, Change from Baseline to 6 Months
  Isokinetic peak torque in Newton-meters of ankle dorsiflexion and plantar flexion (calf muscle) will be obtained using the Biodex Dynamometer. Participants will be seated in a chair tilted slightly back with the right leg elevated resting on a support and right foot strapped to a pedal. The right foot is flexed and extended to move the pedal and obtain the measurements. Three trials of one rep will be done at a speed of 60˚/sec with a one-minute rest in between each trial. The highest torque from the three trials will be used in analysis.
  The change in highest torque in Newton-meters from baseline to intervention completion (3 months) will be used to test the effect of the intervention. The change in highest torque from baseline to follow-up (6 months) will be used to test the persistent effect of the intervention.

SECONDARY OUTCOMES:
Jump Power | Change from Baseline to 3 Months, Change from Baseline to 6 Months
  Jump Power generated from a two-leg counter movement jump will be obtained using the Leonardo Ground Reaction Force Plate (Stratec). The jump motion is recorded using mechanography software. Peak power in kilowatts is obtained. Participants will stand on the plate device and are asked to jump as high as possible by bending the knees and then propelling up. A member of the research team will assist the participant if needed to insure there are no falls. The highest peak power from the 3 jumps will be used in data analysis.
  The change in peak power from baseline to intervention completion (3 months) will be used to test the effect of the intervention. The change in peak power from baseline to follow-up (6 months) will be used to test the persistent effect of the intervention.
Timed up-and-go test | Change from Baseline to 3 Months, Change from Baseline to 6 Months
  The participant sits upright on a stable chair with arm rests (45 cm height) and is allowed to use arms and armrest or the usual walking aid to rise, walk 3 meters to a visible finish line on the floor, turn around, walk back to the chair and sit.
  Time is measured from start to returning to the sitting position with a stop watch to the nearest tenth of a second. The change in the timed up-an-go test from baseline to intervention completion (3 months) will be used to test the effect of the intervention. The change from baseline to follow-up (6 months) will be used to test the persistent effect of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Bonny Specker, Ph.D., Study Director — South Dakota State University

IPD SHARING:
Plan to Share IPD: No